CLINICAL TRIAL: NCT06743087
Title: Effect of Elbow Flexors Fatigue on Hand Grip Strength
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omar Ahmed Hasan Al Askary, Principle investigator, Cairo University
Other Study IDs: P.T.REC/012/005454
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Hand Grip Strength
Keywords: Hand grip strength; Elbow flexors; fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Jamar handheld dynamometer — Jamar handheld dynamometer

SUMMARY:
This study will be conducted to investigate the effect of elbow flexors fatigue on handgrip strength in physiotherapy students

DETAILED DESCRIPTION:
Physiotherapy students rely heavily on hand function throughout their academic and professional careers. Strong hand grip strength is essential for various tasks, including manual therapy techniques, grasping objects, and maintaining writing posture (Lakshmanan et al., 2024; Butt et al., 2022).

Interestingly, research suggests a close link between handgrip strength and endurance, with weakness in one impacting the other (Butt et al., 2022). This highlights the importance of hand function not only for effective treatment delivery but also for students' academic performanceas studies have shown a correlation between handgrip strength and writing speed (Butt et al., 2022).

However, several aspects of a physiotherapy student's life can contribute to elbow flexor fatigue, potentially compromising hand function. These include prolonged static postures while studying from phones or tablets, holding textbooks, and maintaining writing positions during notetaking (Lakshmanan et al., 2024). These factors, prevalent in student life, are likely to continue and potentially worsen in professional practice, where manual therapy techniques and repetitive movements further strain the elbow flexors (Lakshmanan et al., 2024).

Muscle fatigue is characterized by the inability to sustain the required force or power output during activity, ultimately reducing a muscle's capacity to complete tasks over time at a specific load (Li et al., 2024). This physiological phenomenon is accompanied by a subjective experience of increased tiredness or even exhaustion (Li et al., 2024).

Furthermore, muscle fatigue extends beyond a simple lack of energy, demonstrably impairing physical performance and cognitive function. Studies have revealed that fatigue alters muscle activation patterns, potentially increasing the risk of injuries and even fatalities. Notably, research suggests that lower extremity muscle fatigue specifically affects postural control and dynamic balance in older adults while also hindering exercise performance in young adults (Li et al., 2024).

Understanding the relationship between elbow flexor fatigue and hand grip strength in this population is crucial. By investigating this connection, we can gain valuable insights into optimizing hand function for physiotherapy students. This knowledge can be translated into practical strategies to improve treatment efficacy, prevent injuries, and ultimately enhance student success in both academic and professional settings.

ELIGIBILITY:
Inclusion Criteria:

1. Adult non-athletic physiotherapy students with age range between (18: 25) years old
2. Dominant hand is either the right or the left hand
3. Body mass index between (18.5:24.99) Kg/ m2.(

Exclusion Criteria:

1. Traumatic conditions of the upper limb.
2. Previous orthopedic disorders or neurological deficit of the upper limb.
3. Previous surgery of the upper limbs.
4. Any sensory problems.
5. Neuromuscular disease like multiple sclerosis.
6. Pregnancy.
7. Cancer Patients.
8. Immunodeficiency diseases.
9. Psychological disorders (depression - anxiety).
10. Chronic diseases as (diabetes - hypertension)
11. Participants with hand deformity
12. Participants with specific hand muscles weakness

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-12-17 (Estimated); Primary Completion 2025-02-15 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Hand grip strength | 3 months
  Assessing hand grip strength after induced elbow flexors fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Omar Al Askary, Bacheleor, Principal Investigator — Misr University for Science and Technology; Soheir Shehata, Professor, Study Chair — Cairo univerity; Magda Ramadan, Ass. Professor, Study Director — Cairo University; Ahmed Elhamy, Lecturer, Study Director — Misr University for Science and Technology

IPD SHARING:
Plan to Share IPD: No